CLINICAL TRIAL: NCT02975167
Title: Patient Satisfaction During Outpatient Versus Inpatient Foley Catheter Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Responsible Party: Principal Investigator, Vineet Shrivastava, Maternal Fetal Medine Attending, MemorialCare Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 630-15
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Induction of Labor Affected Fetus / Newborn; Cervical Ripening; Patient Satisfaction
Keywords: Induction of labor; mechanical cervical ripening; patient satisfaction; outpatient; cost savings
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Inpatient (Experimental): Subjects randomized to this group will receive the same intervention as the outpatient group -- cervical ripening with Foley catheter -- but remain within the hospital. Subjects will be asked to complete a survey assessing their fears, opinions, anxiety, satisfaction and hours of sleep before and after the catheter is placed and removed, respectively.
  The intervention: randomization to inpatient cervical ripening
  Interventions: Other: Inpatient Cervical Ripening; Procedure: Foley catheter placement; Behavioral: Pre-Foley Questionnaire; Behavioral: Post-Foley Questionnaire; Procedure: Fetal Non-Stress Test
- Outpatient (Experimental): Subjects randomized to this group will receive the same intervention as the inpatient group -- cervical ripening with Foley catheter -- but will be discharged home. Subjects will be asked to return to the hospital when the catheter falls out or if 24 hours has elapsed. They will be given detailed instructions and provided a 24 hour phone number to call should they have any concerns. Subjects will be asked to complete a survey assessing their fears, opinions, anxiety, satisfaction and hours of sleep before and after the catheter is placed and removed, respectively.
  The intervention: randomization to outpatient cervical ripening
  Interventions: Other: Outpatient Cervical Ripening; Procedure: Foley catheter placement; Behavioral: Pre-Foley Questionnaire; Behavioral: Post-Foley Questionnaire; Procedure: Fetal Non-Stress Test

INTERVENTIONS:
Other: Outpatient Cervical Ripening — The experimental arm of the study will be subjects randomized to the outpatient group. Once randomized, subjects will complete a survey assessing their attitudes, fears, anxiety, satisfaction and expected hours of sleep with outpatient induction of labor. Following placement of the Foley catheter, the subjects will be given detailed instructions for which to return to the hospital, as well as provided a 24 hour phone number to call if they have questions. They will be instructed to return to the hospital once the catheter falls out or if 24 hours has passed since its placement. Upon returning to the hospital, subjects will complete another survey assessing their satisfaction with their induction process.
  Other Names: randomization to outpatient cervical ripening
  Arms: Outpatient
Other: Inpatient Cervical Ripening — Once randomized to this group, subjects will complete a survey assessing their attitudes, fears, anxiety, satisfaction and expected hours of sleep with inpatient induction of labor. Following placement of the Foley catheter, the subjects will undergo normal labor monitoring until their Foley catheter either falls out or is removed at 24 hours. At this time subjects will complete another survey assessing their satisfaction with their induction process.
  Other Names: Randomization to inpatient cervical ripening
  Arms: Inpatient
Procedure: Foley catheter placement — Subjects randomized to both the inpatient and the outpatient arms will receive this intervention following completion of a survey. A Bard(TM) 16G two-way 5cc silicone-coated latex Foley catheter will be placed by a physician-member of the research team using a sterile metal speculum and ring forceps, or by hand, depending on physician preference. Once placed within the cervical canal, the Foley will be filled with 60cc of saline
Behavioral: Pre-Foley Questionnaire — Prior to randomization into inpatient or outpatient arms, all subjects will complete a questionnaire assessing their attitudes, opinions, fears and anxiety regarding induction of labor.
Behavioral: Post-Foley Questionnaire — Following removal of the Foley catheter (either by a physician at 24 hours or spontaneously), all subjects will complete the same questionnaire as prior assessing their attitudes, opinions, fears and anxiety regarding their induction of labor.
Procedure: Fetal Non-Stress Test — Following placement of the Foley catheter, all subjects, regardless of arm they are randomized to, will undergo a 20-minute NST. The NST will be read by a physician-member of the research team. If the NST is considered to be suspicious based on the physician's evaluation, subjects randomized to the outpatient arm will be moved to the inpatient arm, but evaluated as part of the outpatient arm on an intent-to-treat basis. All subjects randomized to the inpatient arm will be placed on continuous fetal heart rate monitoring, regardless of physician evaluation of the NST.

SUMMARY:
Labor induction is one of the most common obstetric procedures performed in the U.S. In 2012, the last year for which data is available, 23.7% of all deliveries were the result of inductions. Labor induction first requires cervical ripening, which can be accomplished by several different methods. Vaginal or oral prostaglandins, extra amniotic saline infusion, osmotic dilators and transcervical Foley catheters are all widely used instruments for pre-induction cervical ripening. The ideal cervical ripening tool is safe for both mother and fetus, incurs low cost, does not require extensive monitoring, and causes minimal maternal discomfort. The Foley catheter has been found to be both safe and effective, but little is known about patient satisfaction with the device in an in-patient and out-patient setting. The proposed study will investigate patient satisfaction in a randomized controlled trial of in-patient versus out-patient use of Foley catheters.

DETAILED DESCRIPTION:
Labor induction is one of the most common obstetric procedures performed in the U.S. In 2013, the last year for which data is available, 23.1% of all deliveries were the result of inductions. Labor induction often first requires cervical ripening, which can be accomplished by several different methods.

Pharmacologic cervical ripening approaches include vaginal or oral prostaglandin administration. Mechanical cervical ripening methods include osmotic dilators such as laminaria, and transcervical Foley catheters with or without extra amniotic saline infusion. The ideal cervical ripening tool is effective, safe for both mother and fetus, incurs low cost, does not require extensive monitoring, and causes minimal maternal discomfort.

Several recent meta-analyses have demonstrated both the safety and efficacy of the Foley catheter for pre-induction cervical ripening. When compared to prostaglandins, studies have shown that use of the transcervical Foley catheter for pre-induction cervical ripening results in either shortened or no statistically significant difference in vaginal delivery rates at 24 hours. No studies have demonstrated longer duration to vaginal delivery and cesarean delivery rates are equivalent. In addition, women with Foley catheters experience less uterine hyper-stimulation resulting in fetal heart rate changes as compared to those who receive prostaglandins. Other than one study suggesting increased risks of chorioamnionitis and neonatal infection, the vast majority of research suggests Foley catheters are overwhelming safe with little risk of severe maternal or neonatal morbidity.

Due to its safety profile and the ongoing desire to reduce healthcare costs, many institutions have initiated outpatient cervical ripening protocols. Studies suggest that outpatient cervical ripening with transcervical Foley catheter is both safe and effective. In addition, some studies demonstrate women who underwent outpatient cervical ripening spent less time in the hospital during their labor induction, sometimes resulting in significant cost savings at those institutions. The combination of safety, ease of use and cost savings potential make outpatient cervical ripening with a Foley catheter an appealing tool for both clinicians and patients. However, data on patient satisfaction with almost all methods of cervical ripening is sparse. Existing data on patient satisfaction of outpatient versus inpatient induction of labor stems from prior studies which used vaginal misoprostol gel or isosorbide mononitrate as induction agents. While one study suggests overall satisfaction with outpatient Foley catheter cervical ripening, a randomized controlled trial on this topic has yet to be performed.

ELIGIBILITY:
Inclusion Criteria:

* > 18 yo
* Singleton pregnancy
* ≥ 39 weeks gestation
* Vertex presenting fetus

Exclusion Criteria:

* < 18 years of age
* Maternal cardiac disease
* Class C diabetes mellitus or worse (as defined by the White classification system for diabetes in pregnancy)
* Gestational or chronic hypertension
* Active or history of venous thromboembolic disease requiring chemical anticoagulation
* Bleeding disorders
* History of placental abruption during current gestation
* Fetal anomalies
* Intrauterine growth restriction < 5th percentile
* Prior uterine scar
* Vasa or placenta previa
* Active genital herpes
* Non-vertex fetal lie
* Amniotic fluid index (AFI) < 5cm
* Multiple gestation
* (Pre)eclampsia
* Latex allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-11; Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction scores | Through study completion - expected to be one year
  The primary outcome will be the total score on Part A of the survey, giving an overall rating of the patients' experience with treatment. Means and standard deviations of the total score will be calculated and reported by treatment group among nulliparous and multiparous patients separately. To address the main hypothesis, an ANOVA (analysis-of-variance) will be performed on an intention-to-treat basis and the stratum (nulliparous vs multiparous) will be controlled for in the analysis. The mean difference between treatment groups will be calculated and reported with a 95% confidence interval for the population difference. A two-sample t-test will be used to test for a significant difference in overall rating between in-patient versus out-patient treatment groups.

SECONDARY OUTCOMES:
Multiparous versus Nulliparous subjects | Through study completion - expected to be one year
  Mean differences between in-patient and out-patient treatment will be calculated and reported with 95% confidence intervals among nulliparous and multiparous patients separately. An ANOVA test of interaction will be made in order to address whether multiparous patients rate their experience with the Foley catheter differently than do nulliparous patients.

CONTACTS AND LOCATIONS:
Overall Officials: Vineet Shrivastava, MD, Principal Investigator — Faculty
Locations (1):
- Miller Women's and Children's Hospital Long Beach, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin JA, Hamilton BE, Osterman MJ, Curtin SC, Matthews TJ. Births: final data for 2013. Natl Vital Stat Rep. 2015 Jan 15;64(1):1-65. PMID 25603115
- [Background] Gelber S, Sciscione A. Mechanical methods of cervical ripening and labor induction. Clin Obstet Gynecol. 2006 Sep;49(3):642-57. doi: 10.1097/00003081-200609000-00022. PMID 16885669
- [Background] Jozwiak M, Bloemenkamp KW, Kelly AJ, Mol BW, Irion O, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD001233. doi: 10.1002/14651858.CD001233.pub2. PMID 22419277
- [Background] Jozwiak M, ten Eikelder M, Oude Rengerink K, de Groot C, Feitsma H, Spaanderman M, van Pampus M, de Leeuw JW, Mol BW, Bloemenkamp K; PROBAAT Study Group. Foley catheter versus vaginal misoprostol: randomized controlled trial (PROBAAT-M study) and systematic review and meta-analysis of literature. Am J Perinatol. 2014 Feb;31(2):145-56. doi: 10.1055/s-0033-1341573. Epub 2013 Apr 5. PMID 23564065
- [Background] Kandil M, Emarh M, Sayyed T, Masood A. Foley catheter versus intra-vaginal misoprostol for induction of labor in post-term gestations. Arch Gynecol Obstet. 2012 Aug;286(2):303-7. doi: 10.1007/s00404-012-2292-8. Epub 2012 Mar 21. PMID 22434058
- [Background] Sciscione AC, McCullough H, Manley JS, Shlossman PA, Pollock M, Colmorgen GH. A prospective, randomized comparison of Foley catheter insertion versus intracervical prostaglandin E2 gel for preinduction cervical ripening. Am J Obstet Gynecol. 1999 Jan;180(1 Pt 1):55-60. doi: 10.1016/s0002-9378(99)70149-3. PMID 9914578
- [Background] Heinemann J, Gillen G, Sanchez-Ramos L, Kaunitz AM. Do mechanical methods of cervical ripening increase infectious morbidity? A systematic review. Am J Obstet Gynecol. 2008 Aug;199(2):177-87; discussion 187-8. doi: 10.1016/j.ajog.2008.05.005. PMID 18674661
- [Background] McMaster K, Sanchez-Ramos L, Kaunitz AM. Evaluation of a Transcervical Foley Catheter as a Source of Infection: A Systematic Review and Meta-analysis. Obstet Gynecol. 2015 Sep;126(3):539-551. doi: 10.1097/AOG.0000000000001002. PMID 26244535
- [Background] Maslovitz S, Lessing JB, Many A. Complications of trans-cervical Foley catheter for labor induction among 1,083 women. Arch Gynecol Obstet. 2010 Mar;281(3):473-7. doi: 10.1007/s00404-009-1136-7. Epub 2009 Jun 2. PMID 19488776
- [Background] Sciscione AC, Bedder CL, Hoffman MK, Ruhstaller K, Shlossman PA. The timing of adverse events with Foley catheter preinduction cervical ripening; implications for outpatient use. Am J Perinatol. 2014 Oct;31(9):781-6. doi: 10.1055/s-0033-1359718. Epub 2013 Dec 17. PMID 24347259
- [Background] McKenna DS, Duke JM. Effectiveness and infectious morbidity of outpatient cervical ripening with a Foley catheter. J Reprod Med. 2004 Jan;49(1):28-32. PMID 14976792
- [Background] Kelly AJ, Alfirevic Z, Ghosh A. Outpatient versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2013 Nov 12;(11):CD007372. doi: 10.1002/14651858.CD007372.pub3. PMID 24222365
- [Derived] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803